CLINICAL TRIAL: NCT02212067
Title: A Single-centre, Randomised, Double-blind, Multiple-dose, Placebo-controlled, Parallel-group Trial Investigating the Effects of Semaglutide on ß-cell Function in Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Effects of Semaglutide on ß-cell Function in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3635; 2013-002173-22 (EudraCT Number); U1111-1143-1206 (Other: WHO)
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Semaglutide (Experimental): Total of 12 visits
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator): Total of 12 visits
  Interventions: Drug: placebo
- Healthy subjects (No Intervention): Total of 2 visits

INTERVENTIONS:
Drug: semaglutide — Administered subcutaneously (s.c., under the skin) once weekly for 12 weeks.
  Arms: Semaglutide
Drug: placebo — Administered subcutaneously (s.c., under the skin) once weekly for 12 weeks.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the effects of semaglutide on ß-cell function in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64 years (both inclusive) at the time of signing the informed consent
* For subjects with type 2 diabetes:
* Male and female subjects diagnosed with type 2 diabetes
* Treated with diet and exercise and/or metformin monotherapy. Metformin dose should be unchanged in a period of 30 days prior to screening
* Body Mass Index (BMI) between 20.0-35.0 kg/m^2 (both inclusive)
* Glycosylated haemoglobin (HbA1c) between 6.5-9.0 % (both inclusive)
* For healthy control group for graded glucose infusion:
* Healthy male and female subjects
* BMI between 24.0-32.0 kg/m^2 (both inclusive)
* HbA1c less than 6.5 %

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child bearing potential and not using an adequate contraceptive method. Women of child bearing potential must use an effective method of birth control for the duration of the trial and for subjects with type 2 diabetes for 5 weeks following the last dose of semaglutide. Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices), or sexual abstinence or vasectomised partner
* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ disease including: cardiac, pulmonary, gastrointestinal, hepatic, neurologic, renal, genitourinary and endocrine, dermatologic or hematologic
* Use of any prescription or non-prescription medication which could interfere with trial pharmacokinetic or pharmacodynamic results, as judged by the investigator or specifically: a) current treatment with systemic (oral or i.v.) corticosteroids, non-selective betablockers, b) thyroid hormones are not allowed unless the use of these have been stable during the past 2 month prior to screening
* History of drug/chemical substance abuse within 1 year prior to screening, or a positive result in the urine drug test
* History of alcohol abuse within 1 year prior to screening, or a positive result in the alcohol breath test
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2015-05-11 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin concentration time curve from 0 to 10 minutes after a 25 g glucose bolus i.v. infusion (IVGTT,intravenous glucose tolerance test) over 2 minutes | Day -1, day 86
Area under the serum insulin concentration time curve from 10-120 minutes after a 25 g glucose bolus i.v. infusion (IVGTT). | Day -1, day 86

SECONDARY OUTCOMES:
Area under the insulin secretion rate (ISR)-time curve within 0 to 10 min after i.v. glucose challenge | Day -1, day 86
Area under the ISR-time curve within 10 to 120 min after i.v. glucose challenge | Day -1, day 86
24-hour plasma glucose, glucagon, serum insulin, and C-peptide measured as total AUC0-24h during a test day with 3 standardised meals | Day -1, day 85
Area under the insulin secretion rate (ISR)-time curve within 0 to 10 min after i.v. arginine application; ISR will be derived from the C-peptide concentration profile | Day -1, day 86
Area under the ISR curve over the 5-12 mmol/L (90-216 mg/dL) glucose interval; ISR will be derived from the C-peptide concentration profile | Day -1, day 87
Slope of the ISR vs. glucose curve (dose-response relationship) | Day -1, day 87

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Kapitza C, Dahl K, Jacobsen JB, Axelsen MB, Flint A. Effects of semaglutide on beta cell function and glycaemic control in participants with type 2 diabetes: a randomised, double-blind, placebo-controlled trial. Diabetologia. 2017 Aug;60(8):1390-1399. doi: 10.1007/s00125-017-4289-0. Epub 2017 May 19. PMID 28526920
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com